CLINICAL TRIAL: NCT04452890
Title: PASTIS-Trial: Pre-operative Assessment by Sonourethrography Only in Anterior Urethral Strictures: A Prospective Feasibility Trial
Brief Title: Pre-operative Assessment by Sonourethrography Only in Anterior Urethral Strictures.
Acronym: PASTIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BC-06980-ADP
Record Dates: First submitted 2020-06-12; First posted 2020-07-01 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2020-06

CONDITIONS: Anterior Urethral Stricture, Male
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Intervention Model Description: Single center, prospective feasibility trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sonourethrography (Experimental): Ultrasound of the urethra (Sonourethrography - SUG): In this procedure, a Foley catheter is inserted into the top of the urethra and physiological serum is instilled into the urethra while a linear 7.5 MHz ultrasound probe is placed sagitally on the course of the urethra to detect a narrowing of the urethra.
  Interventions: Diagnostic Test: Sonourethrography

INTERVENTIONS:
Diagnostic Test: Sonourethrography — Ultrasound of the urethra.

SUMMARY:
The choice of the best surgical technique for urethral stricture repair depends on the stricture length. Estimating the length of urethral strictures is therefore of utmost importance.

Different clinical studies have proven that SUG has a higher sensitivity to evaluate the length of urethral strictures compared to RUG or VCUG.

The goal of this study is to assess the feasibility of using SUG as single pre-operative assessment tool in patients with suspicion of anterior urethral strictures. In this way, use of RUG and/or VCUG could be omitted in the pre-operative work-up of patients with anterior urethral strictures, thereby avoiding significant radiation load of patients.

DETAILED DESCRIPTION:
Urethral stricture disease (USD) is a medical condition in which a narrowing of the urethral lumen occurs due to pathological fibrosis and cicatrix formation of the urethral mucosa and surrounding spongious tissue (spongiofibrosis). Urethral strictures may occur at any location from the bladder neck to the external urethral meatus and are categorized based on their localisation in anterior strictures (including the urethral meatus, penile urethra and bulbar urethra) and posterior strictures (including the prostatic urethra and membranous urethra). USD is a disease of all ages but the prevalence increases with increasing age since the cumulative risk of having had urethral instrumentation equally increases. All processes that cause urethral trauma may provoke USD. The majority of strictures nowadays is idiopathic or caused by iatrogenic trauma of the urethra.

The pathological narrowing of the urethral lumen can lead to a wide variety of symptoms which ask for specific diagnostic investigations, in which imaging of the urethra plays a central role. Retrograde urethrography (RUG) and voiding cystourethrography (VCUG) are considered to be the gold standard diagnostic investigation techniques for diagnosis of USD.

In both techniques, contrast is instilled in the urethra through the urethral meatus and radiographic imaging is used to visualize the urethra. RUG and VCUG offer the possibility to visualize the urethra completely and to evaluate the number, length and location of urethral strictures. On the other hand, these techniques have some crucial disadvantages. First and foremost, the radiation load of the genitopelvic region in often young patients is inevitable in RUG and VCUG. Secondly, it is impossible to evaluate the degree of spongiofibrosis with radiographic imaging.

In 1988, McAnnich, et al. were the first to describe sonourethrography (SUG) for the diagnosis of anterior urethral strictures in males. In this technique, a Foley catheter is inserted in the urethral meatus and a physiological solution is instilled in the urethra while a linear 7,5 MHz ultrasound probe is placed sagitally over the course of the urethra. SUG is not only able to evaluate the length and localization of a US, but it also enables the investigator to evaluate the grade of spongiofibrosis.

Different strudies have shown that SUG has a higher sensitivity for the measurement of urethral stricture length compared to classical radiographic imaging such as RUG or VCUG. Since the choice of the most adequate surgical technique depends on the length of the urethral stricture, correct estimation of the urethral stricture length is of the utmost importance.

The goal of this study is to evaluate the feasibility of the use of sonourethrography as single diagnostic tool in the pre-operative diagnostic work-up of males with suspicion of anterior urethral strictures. In this way, classic radiographic imaging such as RUG and VCUG could be omitted in these patients, saving them from a significant radiation load.

Fifty patients with penile strictures and fifty patients with bulbar strictures will be included in this study. When 50% of patients (25 penile and 25 bulbar strictures) have completed the study, an interim analysis will be conducted. If this analysis shows that RUG or VCUG can be omitted in 80% or more of patients, the study will be stopped.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older
* Anterior urethral strictures (except for meatal strictures)

Exclusion Criteria:

* Posterior urethral strictures
* Meatal strictures
* History of hypospadias repair
* History of phalloplasty

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only biological males with anterior urethral stricture disease will be included in the study.
Enrollment: 100 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Sonourethrography feasibility: proportion of patients in whom the pre-operative surgical treatment planning was accurate | 2 years
  To evaluate the proportion of patients in whom the pre-operative surgical treatment planning was accurate based on sonourethrography only.

SECONDARY OUTCOMES:
Identification of predictors for failure of treatment planning by sonourethrography by regression analysis. | 2 years
  To evaluate which factors are predictive for failure of treatment planning by sonourethrography only.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Urology, Ghent University Hospital, Ghent, Belgium